CLINICAL TRIAL: NCT03777150
Title: Is There a Benefit of Postoperative ICU Management After Elective Surgery in Terms of Patient's Outcome, Length of Hospital Stay, Complications and Cost?
Brief Title: Is There a Benefit of Postoperative ICU Management After Elective Surgery in Critical Ill Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Georgia Micha, Anesthesiologist,MD, PhD Principal Investigator, Saint Savvas Anticancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICU postoperative care
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Care; Intensive Care
Keywords: Intensive care; postoperative care; elective surgery
MeSH Terms: interventions — Postoperative Care; Intensive Care Units

STUDY DESIGN:
Intervention Model Description: Group I: admitted into the ICU for postoperative care Group II: admitted into a standard ward for postoperative care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ICU (Experimental): Group ICU:patients are admitted directly into the ICU for postoperative care
  Interventions: Other: Postoperative care in Intensive care unit (ICU)
- Group Ward (Experimental): Group Ward:patients are admitted directly into the standard ward for postoperative care
  Interventions: Other: Postoperative care in standard ward

INTERVENTIONS:
Other: Postoperative care in Intensive care unit (ICU) — Postoperative care in Intensive care unit (ICU)
  Arms: Group ICU
Other: Postoperative care in standard ward — Postoperative care in standard ward
  Arms: Group Ward

SUMMARY:
Postoperative care of high risk patients in the Intensive Care Unit (ICU) has for long been considered to be the gold standard of care in terms of reducing perioperative mortality.New evidence from a 7-day cohort study involving 27 countries comes to question this practice. The primary objective of our study is to detect any benefit of postoperative ICU care after elective surgery in terms of patient's outcome, length of hospital stay, complications and cost.

DETAILED DESCRIPTION:
A prospective analysis of high perioperative risk patients that are about to be subjected into an elective operation will be included into the study. They will be allocated into two groups. Group ICU patients are those that are admitted into the ICU for postoperative care and those that are admitted into a standard ward consist Group Ward. Demographic data, the length of hospital stay, the outcome, the need of mechanical ventilation, the complications and the total cost will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients that will be scheduled for an elective operation and are considered to be in a high perioperative risk

Exclusion Criteria:

* Patients that are operated on an emergency basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total length of hospital stay | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  The total length of patient's hospital stay will be recorded

SECONDARY OUTCOMES:
Preoperative length of hospital stay | From date of hospital admission until the date of operation or date of death from any cause, whichever came first, assessed up to 6 months
  The preoperative length of patient's hospital stay will be recorded
Postoperative length of hospital stay | From date of surgical operation until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  The postoperative length of patient's hospital stay will be recorded
Postoperative complications | From date of surgical operation until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  All postoperative complications will be recorded
Patient's outcome at 28 days postoperatively | From the first postoperative day until 28 days postoperatively
  28 day postoperative mortality will be recorded
Total cost of hospital care | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  The total cost of hospital care will be recorded for every patient
Postoperative cost of hospital care | From date of surgical operation until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  The postoperative cost of hospital care will be recorded for every patient

CONTACTS AND LOCATIONS:
Overall Officials: Anna Efthimiou, Head of the department, Study Director — Saint Savvas Anticancer hospital of Athens
Locations (1):
- Saint Savvas Anticancer Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided